CLINICAL TRIAL: NCT04578262
Title: Epley Manoeuvre for Posterior Semi-circular Canal Benign Paroxysmal Positional Vertigo in People With Multiple Sclerosis: Protocol of a Randomized Controlled Trial
Brief Title: Epley Manoeuvre in Participants With Multiple Sclerosis Diagnosed From Benign Paroxysmal Positional Vertigo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Cristina García Muñoz, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Seville Protocol
Record Dates: First submitted 2020-09-20; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Benign Paroxysmal Positional Vertigo; Multiple Sclerosis
Keywords: Multiple Sclerosis; Benign Paroxysmal Positional Vertigo; Epley Manoeuvre; Vertigo; Dizziness
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Multiple Sclerosis; Vertigo; Dizziness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epley Manoeuvre (Experimental): Epley manoeuvre in participants with Multiple Sclerosis who suffer from benign paroxysmal positional vertigo. Only one administration.
  Interventions: Procedure: Epley Manoeuvre
- Sham Manoeuvre (Sham Comparator): The second group will received a sham manoeuvre. However after the experimental intervention ends, this groups will also receive Epley manoeuvre.
  Interventions: Procedure: Sham Manoeuvre

INTERVENTIONS:
Procedure: Epley Manoeuvre — This manoeuvre is constituted by five steps. In the first step, while the patient is in supine posture the head will be positioned 45 degrees turned towards the unaffected ear and the head slightly overhang on the edge of the couch. In this second step maintaining the previous position of the head, physiotherapist will turn head 45 degrees turned towards the affected ear. Next, in the third step, the whole body will turn until is located 135 degrees from the baseline supine position. In the fourth step, while the head keeps turned to the affected ear the subject will be incorporated until he is sitting. In the fifth step, while the subject is seated with the head in neutral position the chin will be bended 20 degrees. Each procedure will be held among 30 seconds or two minutes, while the dizziness or the nystagmus vanish. The intervention will be conducted at the Physical Therapy Department of the University of Sevilla (Spain).
  Other Names: canalith repositioning procedure for posterior semi-circular canal
  Arms: Epley Manoeuvre
Procedure: Sham Manoeuvre — The sham manoeuvre consist is going to star with the participant in a neutral seated position. Sum to it, head is rotated 45 degrees towards the unaffected vestibule. After that, the participant will be guided by the physiotherapist to a lateral decubitus position towards the affected side on which his nose will be pointing above. To conclude, the seated position will be reached again without head rotation. Each position of the sham manoeuvre will be maintained along one minute. During all the process the videonystagmography glasses will be dressed by participants and they will be indicated not to close eyes in the intervention. After the execution of the manoeuvre, also this group will be evaluated 48 hours after. The intervention will be conducted at the Physical Therapy Department of the University of Sevilla (Spain).
  Arms: Sham Manoeuvre

SUMMARY:
Vertigo, dizziness and control postural disturbance are one of the most disabling symptoms in Multiple Sclerosis. These could be caused by a peripheral or central vestibular disorder. Although, central vestibular damage is more prevalent, peripheral vestibular disturbance aetiology is significantly common in this disease. Within peripheral vestibulopathy, benign paroxysmal positional vertigo is the most common syndrome. Impairments of posterior semi-circular canals in benign paroxysmal positional vertigo represent among the 60-90 % of the cases. Gold standard treatment in this syndrome is the canalith repositioning procedure, called Epley manoeuvre. This manoeuvre has been deeply investigated in previous studies for participants who only suffer from benign paroxysmal positional vertigo. Any randomized clinical trials have been carried out to assess the effectiveness of Epley manoeuvre. However, a retrospective research and a case study reported encouraging results for the resolution of posterior semi-circular canal benign paroxysmal positional vertigo, through the Epley manoeuvre. The main objective of the study is to assess the effectiveness of the Epley Manoeuvre for the improvement of the benign paroxysmal positional vertigo of participants with multiple sclerosis, compared to a passive control group.

DETAILED DESCRIPTION:
After given oral and written information to participants, they will be freedom to decide their wish to participate. After the invitation, those participants who desire to be part of study will sign the written informed consent.The study describes a two-arms, parallel groups design and double-blind randomized clinical trial. A prospective study with randomized and conceal allocation will be performed to prevent possible bias. Participants and evaluators will be blinded to group allocation. The randomized controlled trial have 3 evaluations of the sample, that will be carried out at baseline, immediately after intervention and 48 hours later

ELIGIBILITY:
Inclusion Criteria:

* Adults of both genders aged from 18 to 65 years old.
* clinically diagnosed of any MS subtype (relapsing-remitting, primary progressive and secondary progressive),
* with an Expanded Disability Status Scale (EDSS) ranging from 1 to 5 points,
* diagnosed of posterior semi-circular canals benign paroxysmal positional vertigo by an otolaryngologist and a physical therapist expert in vestibular rehabilitation.

Exclusion Criteria:

* Changes in MS pharmacotherapy within the last 3 months,
* BPPV treatments as vestibular sedatives, corticosteroids, morphic and antihistamines, at least 72 hours before intervention,
* alcohol consumption in the last 72 hours,
* severe visual impairments,
* participants who have received vestibular rehabilitation within the last 3 months,
* existence of any other neurologic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Changes in the conversion of a positive to a negative Dix Hallpike Test | Baseline, immediately after intervention and 48 hours after intervention.
  The performance of Dix Hallpike Test consists on a participant sit on a table and the head is turn 45 degrees towards the tested side. Once this position is stablished, the evaluator is going to laid back the participant in a quick movement sum to a neck extension of 20 degrees with the affected ear down. Throughout the process subject will be indicated to keep eyes open to allow the search of nystagmus. If torsional nystagmus or vertigo appears while the head is down it is indicative of posterior canal benign paroxysmal positional vertigo.

SECONDARY OUTCOMES:
Impact of dizziness in the quality of life in participants with Multiple Sclerosis. Dizziness Handicap Inventory (DHI). | Baseline, immediately after intervention and 48 hours after intervention.
  Dizziness Handicap Inventory is a self-assessment questionnaire of 25- items and the total score is 100. The score is calculated by summing ordinal scales responses, higher scores means higher level of disability and handicap constituted by the physical, emotional and functional subscale. Physical and emotional subscales range from 0 to 36 points, and functional from 0 to 28.
Independency in activities of daily living measure by Vestibular Disorders Activities of Daily Living Scale (VADL). | Baseline, immediately after intervention and 48 hours after intervention.
  Vestibular Disorders Activities of Daily Living Scale (VADL) is a self-reported questionnaire that measures the independence on activities of daily living in people with vestibular disorders. This scale is composed by 28 items divided in three subcategories: 12 questions of functional skills, 9 questions of ambulation skills and 7 questions of instrumental skills. Each item is rate un a 10-point scale, in which higher score means less independence in ADL. The total score is the median of each subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina García-Muñoz, Principal Investigator — University of Seville; Maria Jesus Casuso-Holgado, Principal Investigator — University of Seville; Marilo Dolores Cortes-Vega, Principal Investigator — University of Seville

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Garcia-Munoz C, Cortes-Vega MD, Hernandez-Rodriguez JC, Palomo-Carrion R, Martin-Valero R, Casuso-Holgado MJ. Epley manoeuvre for posterior semicircular canal benign paroxysmal positional vertigo in people with multiple sclerosis: protocol of a randomised controlled trial. BMJ Open. 2021 Mar 18;11(3):e046510. doi: 10.1136/bmjopen-2020-046510. PMID 33737443